CLINICAL TRIAL: NCT00006501
Title: The Prevalence and Prognostic Significance of T Wave Alternans in Patients With Severe Congestive Heart Failture
Brief Title: Prognostic Significance of T Wave Alternans
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAAB1399; R01HL064862 (NIH)
Record Dates: First submitted 2000-11-16; First posted 2000-11-17 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Heart Diseases; Ventricular Arrhythmia; Ventricular Fibrillation; Death, Sudden, Cardiac; Heart Arrest
MeSH Terms: conditions — Heart Diseases; Ventricular Fibrillation; Death, Sudden, Cardiac; Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ECG recording: After the tests are completed, people who enroll in this study are followed by telephone, 1, 4, 8, 12 16, 20 and 24 months. During these follow-up telephone calls a research coordinator asks about the participant's health condition and about cardiovascular medications that are being taken.
  Interventions: Procedure: ECG

INTERVENTIONS:
Procedure: ECG — A diagnostic tool that is routinely used to assess the electrical and muscular functions of the heart (non-experimental).
  Other Names: Electrocardiogram

SUMMARY:
To evaluate whether T Wave Alternans can predict ventricular arrhythmias and sudden cardiac death (SCD) in a prospective epidemiologic natural history study.

The prospective epidemiologic pilot study included 550 patients that had left ventricular dysfunction and no history of sustained ventricular arrhythmias. The primary hypothesis tested was whether there was an increased risk of having an arrhythmic event when T Wave Alternans was present in the patient. The secondary aims included comparing risk due to T Wave Alternans between the ischemic patients and non-ischemic patients and assessing whether T Wave Alternans remained an independent predictor of risk upon adjustment for other known risk factors for arrhythmic events such as ejection fraction, ventricular ectopy, NSVT, average NN interval, and RR interval variability.

The study approach was a standard epidemiologic surveillance technique. The subject population consisted of individuals with Class I to III heart failure who will underwent a TWA and Holter monitor test and then were followed for up to two years or until arrhythmic events occured.

DETAILED DESCRIPTION:
Sudden cardiac death accounts for approximately 400,000 deaths each year in the United States and remains a health problem of epidemic proportions. Most sudden cardiac deaths are caused by fatal ventricular arrhythmias. An effort aimed at the primary prevention of sudden cardiac death requires efficient identification of patients who are at high enough risk for having these arrhythmias to warrant aggressive prophylactic therapy. A number of recently completed, randomized clinical trials have demonstrated that an implantable cardiac defibrillator (ICD) can prevent sudden cardiac death in a highly selected group of high-risk patients. When these trials are viewed together, the only patients in whom the prophylactic implantation of an ICD has proven benefit are those patients identified by documented, spontaneous or inducible, sustained ventricular arrhythmias.

Two randomized treatment trials (MADIT II, SCD-HEFT) tested the hypothesis that implantation of an ICD would reduce mortality in patients with congestive heart failure (CHF) and left ventricular dysfunction without any further risk tratification. However, the implications of these two trials-implantation of an ICD in every patient with CHF-were unlikely to be accepted either by the medical community or by health care payers. More efficient methods of risk stratification were necessary to identify those patients with CHF who were most likely to benefit from prophylactic treatment with an ICD.

T Wave Alternans is a subtle every-other-beat variation in electrocardiographic T waves that is prognostic of patients at high risk for life-threatening cardiac arrhythmias and sudden cardiac death. It has recently been shown that T Wave Alternans (TWA) measured during exercise is strongly associated with inducible monomorphic CVT and with subsequent spontaneous arrhythmic events. This preliminary data suggest that TWA may be an efficient and non-invasive surrogate for electrophysiologic testing to screen patients who may be at high-risk for sudden cardiac death.

ELIGIBILITY:
Inclusion Criteria

1. Patients with left ventricular dusfunction
2. Patients with non-ischemic cardiomyopathy

Exclusion Criteria

1. Patients not at high risk for sudden cardiac death (SCD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with left ventricular dusfunction or non-ischemic cardiomyopathy, and are at high risk for sudden cardiac death.
Sampling Method: Non-Probability Sample
Enrollment: 549 (Actual)
Dates: Start 2003-01; Primary Completion 2009-12 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Pevalence of SCD with earlier testing that indicated TWA | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: John Bigger, Principal Investigator — Professor Emeritus of Medicine and Pharmacology, Columbia University; John Bigger, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

REFERENCES:
- [Background] Bloomfield DM, Bigger JT, Steinman RC, Namerow PB, Parides MK, Curtis AB, Kaufman ES, Davidenko JM, Shinn TS, Fontaine JM. Microvolt T-wave alternans and the risk of death or sustained ventricular arrhythmias in patients with left ventricular dysfunction. J Am Coll Cardiol. 2006 Jan 17;47(2):456-63. doi: 10.1016/j.jacc.2005.11.026. Epub 2005 Dec 15. PMID 16412877